CLINICAL TRIAL: NCT01532999
Title: A Multisite Randomized Controlled Trial of Mindfulness Meditation Therapy for PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPLE-004-11S
Record Dates: First submitted 2011-12-08; First posted 2012-02-15 (Estimated); Results first posted 2015-04-08 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Posttraumatic Stress Disorder; Meditation; Present Centered Group Therapy; mindfulness; MBSR; complementary alternative medicine
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mindfulness Based Stress Reduction (Experimental): Mindfulness Based Stress Reduction (MBSR) is a manualized program involving 8 weekly classes and a single 6-hour silent retreat session based on a systematic procedure to develop enhanced non-reactive awareness of the moment-to-moment experience of perceptible mental processes.
  Interventions: Behavioral: Mindfulness Based Stress Reduction
- Present Centered Group Therapy (Sham Comparator): Present Centered Group Therapy (PCGT) serves as a credible control for the nonspecific effects of a group-based intervention (i.e. controls for time, attention, expectation of recovery, and recognition of the illness).
  Interventions: Behavioral: Present Centered Group Therapy

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction — MBSR is a manualized program involving 8 weekly classes and a single 6-hour silent retreat session based on a systematic procedure to develop enhanced non-reactive awareness of the moment-to-moment experience of perceptible mental processes.
  Other Names: MBSR
  Arms: Mindfulness Based Stress Reduction
Behavioral: Present Centered Group Therapy — The comparison control group will be PCGT, which was initially developed for use as a control group in a VA multi-site study that tested the effects of Trauma-Focused Group Therapy. Correspondingly, PCGT serves as a credible control for the nonspecific effects of a group-based intervention (i.e. controls for time, attention, expectation of recovery, and recognition of the illness).
  Other Names: PCGT
  Arms: Present Centered Group Therapy

SUMMARY:
Currently, veterans with posttraumatic stress disorder (PTSD) are typically treated with antidepressants which have limited efficacy and yield extremely low remission rates. New and improved treatments are sorely needed, especially in light of the inadequate evidence to support the efficacy of most pharmacologic and most psychotherapy treatments for PTSD. Complementary and Alternative Medicine practices, such as meditation, may fill this void. Several other illnesses often found in association with PTSD, such as chronic pain, anxiety, and depression, have shown positive response to meditation, specifically Mindfulness Based Stress Reduction (MBSR). MBSR is manualized program involving 8 weekly classes and a single 6-hour silent retreat session based on a systematic procedure to develop enhanced non-reactive awareness of the moment-to-moment experience of perceptible mental processes. MBSR is well tolerated, already well disseminated. MBSR has been shown to be effective in reducing conditions that are commonly associated with PTSD, including pain, depression, anxiety and panic, and insomnia. The investigators are conducting a multisite study of Mindfulness Based Stress Reduction (MBSR) compared to Present Centered Group Therapy (PCGT) for the treatment of PTSD. The primary aim of this study will be to determine how well the MBSR form of meditation, i.e. MBSR, works to treat symptoms of PTSD in veterans compared to PCGT. The investigators will evaluate the effects of treatment on levels of mindfulness, depression, PTSD symptom clusters, and response rates. The investigators will evaluate veterans' satisfaction and acceptability of the MBSR intervention. Additionally, biomarkers will be utilized to aid in our understanding of the pathophysiology of meditation and explore the relationship between treatment outcome and neuroimmune response.

DETAILED DESCRIPTION:
This study is a prospective, randomized (1:1), controlled multisite study of MBSR in 180 veterans with PTSD. The investigators will compare the clinical outcomes of MBSR to a credible group therapy control condition called Present Centered Group Therapy (PCGT). The investigators will to evaluate the efficacy of MBSR in the treatment of PTSD, as defined by the Clinician Administered PTSD Scale (CAPS), a gold standard measure that is clinically relevant to PTSD. The CAPS will be rated by a trained assessor who is blind to the whether or not the participant receives the MBSR or PCGT intervention. Secondarily, the investigators will evaluate the effects of MBSR on mindfulness, depression, PTSD symptom clusters, rates of response and evaluate the safety and tolerability of MBRS. The investigators will also explore the subjects' acceptance of and satisfaction with MBSR, whether or not the subjects' treatment preference influences outcome; the stress-immunological-biomarkers as they relate to treatment outcome; and the durability of therapeutic effects of MBSR in the treatment of PTSD.

Study Design Overview: Male and female subjects from Active Duty, Reserves, National Guard and/or Veterans with a diagnosis of PTSD will be prospectively randomized 1:1 to receive either MBSR Group therapy or Present Centered Therapy (PCGT) Group (control) for 8 weeks. A cluster of at least 12 participants will be randomized individually to either MBRS or PCGT group therapies, which results in at least 6 participants in each intervention group. A total of 30 groups (15 MBSR Groups and 15 PCGT Groups) are anticipated across three clinical research sites involving at least three different MBSR and three different PCGT instructors/therapists. Outcome assessments (single-blind CAPS and self-report measures) will be obtained at baseline, week 3, week 6, and week 9 (primary endpoint). These assessments will be repeated post-acute treatment at week 16 as an exploratory measure of short-term durability effects.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization form.
* > or = 18 years of age.
* Diagnosis of PTSD (DSM-IV-TR criteria; confirmed by MINI and CAPS).
* Total CAPS score > 45 for the week prior to randomization.
* No substance use disorders (except for nicotine, caffeine) for 2 weeks prior to randomization (Able to Travel to the clinical sites in Tuscaloosa, AL, Atlanta, GA, or Charleston, SC

Exclusion Criteria:

* Lifetime history of bipolar I, schizophrenia, schizoaffective or cognitive disorders (MINI)
* Actively considering plans of suicide or homicide (assessed by clinical interview)
* Psychotic symptoms that in the investigator's opinion impair the subject's ability to give informed consent and participate in the study interventions
* Severe cognitive disorder (Dementia, severe Traumatic Brain Injury)
* Clinically significant unstable or severe medical condition that would contraindicate study participation or expose them to an undue risk of a significant adverse event.
* In regard to vulnerable patient populations, persons with dementia, minors (<age 19), the elderly (>age 65), prisoners and the terminally ill are excluded.
* Individuals with significant psychotic or dissociative symptoms or severe personality disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2012-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori L Davis, MD AB, Principal Investigator — Tuscaloosa VA Medical Center, Tuscaloosa, AL
Locations (3):
- United States (3):
  - Tuscaloosa VA Medical Center, Tuscaloosa, AL, Tuscaloosa, Alabama
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina

REFERENCES:
- [Derived] Shapira I, Richman J, Pace TWW, Lim KO, Polusny MA, Hamner MB, Bremner JD, Mumba MN, Jacobs ML, Pilkinton P, Davis LL. Biomarker Response to Mindfulness Intervention in Veterans Diagnosed with Post-traumatic Stress Disorder. Mindfulness (N Y). 2022 Oct;13(10):2448-2460. doi: 10.1007/s12671-022-01969-6. Epub 2022 Sep 12. PMID 36938380

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 254 participants signed informed consent; 214 participants were randomized; and 191 randomized participants attended at least one MBSR or PCGT session and were included in the modified intent-to-treat analysis for which results are displayed.
Period: Overall Study
Arm/Group | Mindfulness Based Stress Reduction | Present Centered Group Therapy
Started | 96 | 95
Completed | 65 | 77
Not Completed | 31 | 18
Not completed — Lost to Follow-up | 14 | 8
Not completed — Physician Decision | 1 | 2
Not completed — Withdrawal by Subject | 5 | 0
Not completed — Relocated | 2 | 0
Not completed — should not have been randomized | 1 | 0
Not completed — substantial noncompliance | 2 | 0
Not completed — no show for week 9 assessments | 6 | 4
Not completed — Adverse Event | 0 | 1
Not completed — incarcerated | 0 | 1
Not completed — New job | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness Based Stress Reduction | Present Centered Group Therapy | Total
Number analyzed (Participants) | 96 | 95 | 191
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (11) | 51 (8.3) | 51 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31
  Male | 80 | 80 | 160
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 63 | 59 | 122
  White | 30 | 31 | 61
  More than one race | 3 | 3 | 6
  Unknown or Not Reported | 0 | 2 | 2
CAPS Total [Mean (Standard Deviation); unit: units on a scale] — Clinician Administered PTSD Scale (CAPS) is a 17-item standard rating scale that measures PTSD severity with scores ranging from 0-136 (higher score = more severe). Scores of frequency and intensity are summed for the 17-items to yield the total CAPS score.
  units on a scale | 84.3 (19.5) | 80.7 (16.7) | 83 (18.2)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Clinician Administered PTSD Scale
Description: Clinician Administered PTSD Scale (CAPS) is a 17-item standard rating scale that measures PTSD severity with scores ranging from 0-136 (higher score = more severe). Scores of frequency and intensity are summed for the 17-items to yield the total CAPS score.
Time Frame: Baseline to week 9
Population: All participants who were randomized and attended at least one intervention session.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness Based Stress Reduction | Present Centered Group Therapy
Number analyzed (Participants) | 96 | 95
units on a scale | -22.4 (27) | -15.9 (22.9)
Statistical Analysis 1: Comparison: Mindfulness Based Stress Reduction vs Present Centered Group Therapy; Three-level mixed-effects linear regression analysis comparing MBSR and PCGT groups over 9 weeks. Data structure involved repeated measures over time nested within participant, who in turn, was nested within a therapy group. Models included a random intercept, a random slope, and fixed effects for treatment condition, time, and the stratification variable (site). Rejection of the null hypothesis of no treatment effect if this interaction was statistically significant (two-tailed α = .05); Test type: Superiority or Other; p = 0.5, Regression, Linear

2. Secondary Outcome: Change From Baseline in PTSD Checklist (PCL)
Description: PTSD Checklist (PCL) is a 17-item self-report scale intended to measure PTSD symptom severity. The PCL has demonstrated excellent internal consistency (alpha = .94-.97), and test-retest reliability over 2 to 3 days was .96 for Vietnam veterans. Respondents rate each item from 1 ("not at all") to 5 ("extremely") to indicate the degree to which they have been bothered by that particular symptom over the past month. Thus, total possible scores (items summed) range from 17 to 85 (higher score is more severe). A cut-off score of 50 indicates a probable diagnosis of PTSD.
Time Frame: Baseline to week 9
Population: All participants who were randomized and attended at least one intervention session.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness Based Stress Reduction | Present Centered Group Therapy
Number analyzed (Participants) | 96 | 95
units on a scale | -8.6 (15.8) | -6.7 (12)
Statistical Analysis 1: Comparison: Mindfulness Based Stress Reduction vs Present Centered Group Therapy; Three-level mixed-effects linear regression analysis comparing MBSR and PCGT groups over 9 weeks; Test type: Superiority or Other; p = 0.57, Regression, Linear

3. Secondary Outcome: Change From Baseline in Five Facet Mindfulness Questionnaire (FFMQ)
Description: Five Facet Mindfulness Questionnaire (FFMQ) is used to evaluate the effects of MBSR vs. PCGT on mindfulness (S1). The FFMQ is a 39-item self-report instrument that assesses the general tendency to be mindful in daily life through 5 facets: observing, describing, acting with awareness, non-judging of inner experience, non-reactivity to inner experience. Increases in FFMQ mediate improvements in well being in observational studies of MBSR. Each item is rated 1 to 5 ("never or very rarely true" to "very often or always true"). Some of the items are reverse scored (R). Scoring Information: Observe items:1, 6, 11, 15, 20, 26, 31, 36; Describe items: 2, 7, 12R, 16R, 22R, 27, 32, 37; Act with Awareness items: 5R, 8R, 13R, 18R, 23R, 28R, 34R, 38R; Nonjudge items: 3R, 10R, 14R, 17R, 25R, 30R, 35R, 39R; Nonreact items: 4, 9, 19, 21, 24, 29, 33. Total all subscales for score (higher score = greater degree of mindfulness). Score range 39-195 with higher=more mindfulness.
Time Frame: Baseline to week 9
Population: All participants who were randomized and attended at least one intervention session.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness Based Stress Reduction | Present Centered Group Therapy
Number analyzed (Participants) | 96 | 95
units on a scale | 5.2 (16.6) | 2.1 (13.2)

4. Secondary Outcome: Change From Baseline in Patient Health Questionnaire (PHQ-9)
Description: Patient Health Questionnaire (PHQ-9) is a brief 9-item measure of depressive symptoms that has established reliability and validity in community and clinical populations. All items are summed for total score ranging from 0 to 27 (higher score = more severe depression).
Time Frame: Baseline to week 9
Population: All participants who were randomized and attended at least one intervention session.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness Based Stress Reduction | Present Centered Group Therapy
Number analyzed (Participants) | 96 | 95
units on a scale | -3.2 (6.6) | -1.6 (6.3)
Statistical Analysis 1: Comparison: Mindfulness Based Stress Reduction vs Present Centered Group Therapy; Three-level mixed-effects linear regression analysis comparing MBSR and PCGT groups over 9 weeks; Test type: Superiority or Other; p = 0.4, Regression, Linear

5. Secondary Outcome: Change From Baseline in CAPS B Subscale
Description: Clinician Administered PTSD Scale (CAPS) B subscale measures the re-experiencing cluster (i.e. B criterion) of PTSD symptoms and includes the first 5 items of the CAPS, which is a clinician-administered assessment of posttraumatic stress disorder (PTSD) symptoms. Frequency and intensity scores for each item is summed for a range of 0 to 40 (higher score = more severe PTSD).
Time Frame: Baseline to week 9
Population: All participants who were randomized and attended at least one intervention session.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness Based Stress Reduction | Present Centered Group Therapy
Number analyzed (Participants) | 96 | 95
units on a scale | -7.7 (10.4) | -6.2 (8.9)
Statistical Analysis 1: Comparison: Mindfulness Based Stress Reduction vs Present Centered Group Therapy; Three-level mixed-effects linear regression analysis comparing MBSR and PCGT groups over 9 weeks; Test type: Superiority or Other; p = 0.8, Regression, Linear

6. Secondary Outcome: Change From Baseline in CAPS C Subscale
Description: Clinician Administered PTSD Scale (CAPS) C subscale measures the avoidance and emotional numbing cluster (i.e. C criterion) of PTSD symptoms and includes the items 6 - 12 items of the CAPS, which is a clinician-administered assessment of posttraumatic stress disorder (PTSD) symptoms. Frequency and intensity scores for each item is summed for a range of 0 to 56 (higher score = more severe PTSD).
Time Frame: Baseline to week 9
Population: All participants who were randomized and attended at least one intervention session.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness Based Stress Reduction | Present Centered Group Therapy
Number analyzed (Participants) | 96 | 95
units on a scale | -8.8 (12.6) | -6.8 (10.8)
Statistical Analysis 1: Comparison: Mindfulness Based Stress Reduction vs Present Centered Group Therapy; Three-level mixed-effects linear regression analysis comparing MBSR and PCGT groups over 9 weeks; Test type: Superiority or Other; p = 0.4, Regression, Linear

7. Secondary Outcome: Change From Baseline in CAPS D Subscale
Description: Clinician Administered PTSD Scale (CAPS) D subscale measures the hyperarousal cluster (i.e. D criterion) of PTSD symptoms and includes the items 13 - 17 of the CAPS, which is a clinician-administered assessment of posttraumatic stress disorder (PTSD) symptoms. Frequency and intensity scores for each item is summed for a range of 0 to 40 (higher score = more severe PTSD).
Time Frame: Baseline to week 9
Population: All participants who were randomized and attended at least one intervention session.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness Based Stress Reduction | Present Centered Group Therapy
Number analyzed (Participants) | 96 | 95
units on a scale | -5.9 (9.3) | -3 (7.6)
Statistical Analysis 1: Comparison: Mindfulness Based Stress Reduction vs Present Centered Group Therapy; Three-level mixed-effects linear regression analysis comparing MBSR and PCGT groups over 9 weeks; Test type: Superiority or Other; p = 0.35, Regression, Linear

8. Secondary Outcome: PTSD Response
Description: Greater than or equal to 30% improvement on PTSD CAPS scale
Time Frame: Baseline to week 9
Population: All participants who were randomized and attended at least one intervention session.
Measure: Number; unit: percentage of participants
Arm/Group | Mindfulness Based Stress Reduction | Present Centered Group Therapy
Number analyzed (Participants) | 96 | 95
percentage of participants | 45.2 | 37.7
Statistical Analysis 1: Comparison: Mindfulness Based Stress Reduction vs Present Centered Group Therapy; Mixed effects logistic regression analysis; Test type: Superiority or Other; p = 0.3, Regression, Logistic

9. Secondary Outcome: PTSD Remission
Description: Total CAPS score of less than or equal to 45 at week 9 (single observation point)
Time Frame: Week 9
Population: All participants who were randomized and attended at least one intervention session.
Measure: Number; unit: percentage of participants
Arm/Group | Mindfulness Based Stress Reduction | Present Centered Group Therapy
Number analyzed (Participants) | 96 | 95
percentage of participants | 30.7 | 27.3
Statistical Analysis 1: Comparison: Mindfulness Based Stress Reduction vs Present Centered Group Therapy; Mixed effects logistic regression analysis; Test type: Superiority or Other; p = 0.7, Regression, Logistic

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the 17 week follow-up period for each participant.
Arm/Group | Mindfulness Based Stress Reduction | Present Centered Group Therapy
Serious Adverse Events (participants affected / at risk) | 4/96 | 4/95
Other Adverse Events (participants affected / at risk) | 0/96 | 0/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mindfulness Based Stress Reduction (N=96) | Present Centered Group Therapy (N=95)
wisdom tooth infection (Infections and infestations) | 1 (1) | 0 (0) — wisdom tooth infection requiring medical inpatient hospitalization
suicidal and homicidal feelings (Psychiatric disorders) | 3 (3) | 2 (2) — suicidal and homicidal feelings; not related to study or intervention, resulting in psychiatric inpatient admission
Hypotension (Cardiac disorders) | 0 (0) | 1 (1) — Hypotension; preexisting coronary artery disease; unrelated to study or intervention; resulting in medical inpatient hospitalization
swollen scrotum (Reproductive system and breast disorders) | 0 (0) | 1 (1) — medical inpatient hospitalized for swollen scrotum; unrelated to study or intervention

LIMITATIONS AND CAVEATS:
Limitations: PCGT may be more active than originally anticipated and is thus an active control rather than neutral control

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No